CLINICAL TRIAL: NCT02724371
Title: A Study of the Safety and Effectiveness of the Mentor Smooth and Textured Larger Size MemoryGel Ultra High Profile Breast Implants in Subjects Who Are Undergoing Primary Breast Reconstruction or Revision Reconstruction
Brief Title: A Study of the Safety and Effectiveness of the Mentor Larger Size MemoryGel Ultra High Profile Breast Implants in Subjects Who Are Undergoing Primary Breast Reconstruction or Revision Reconstruction
Acronym: Athena
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEN-15-001
Record Dates: First submitted 2016-03-21; First posted 2016-03-31 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Breast Reconstruction, Revision Breast Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary Breast Reconstruction (Experimental): Participants who meet the requirements for primary breast reconstruction (have not had previous silicone or saline breast implants, not including tissue expanders) and have been implanted with Mentor Larger Size MemoryGel Ultra High Profile Breast implants
  Interventions: Device: Mentor Larger Size MemoryGel Ultra High Profile Breast Implant
- Revision Breast Reconstruction (Experimental): participants who meet the requirements for revision breast reconstruction (have had previous silicone or saline breast implants) and have been implanted with Mentor Larger Size MemoryGel Ultra High Profile Breast implants
  Interventions: Device: Mentor Larger Size MemoryGel Ultra High Profile Breast Implant

INTERVENTIONS:
Device: Mentor Larger Size MemoryGel Ultra High Profile Breast Implant — The Mentor smooth and Siltex® larger size MemoryGel® Ultra High Profile (UHP-L) breast implants are large round silicone gel-filled breast implants. The devices are made with cross linked layers of silicone to provide the prosthesis with elasticity and integrity.
  Other Names: UHP-L Breast Implant

SUMMARY:
The study will evaluate the safety and effectiveness with the Mentor MemoryGel® Larger Size Ultra High Profile (UHP-L) Breast Implants.

DETAILED DESCRIPTION:
Subjects, whose body shape is suited to a larger size implant than are currently available, will have their breasts reconstructed using the UHP-L Breast Implants either for the first time after a full mastectomy or as a revision of a previous breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female and is at least 18 years old
* A candidate for:
* Primary breast reconstruction in women at least 18 years old with surgically absent breast tissue (two-stage reconstruction [tissue expanders utilized with or without the use of human acellular dermal matrices (ADM), limited to AlloDerm® and FlexHD® PLIABLE, utilized in a prior surgery to expand tissue for study device placement] to replace breast tissue post-mastectomy)
* Revision surgery in women at least 18 years old with surgically absent breast tissue (previous reconstruction with silicone-filled or saline-filled implants or revision reconstruction requiring expansion surgery prior to surgery for study device implantation, with or without the use of human acellular dermal matrices (ADM), limited to AlloDerm® and FlexHD® PLIABLE, utilized in a prior surgery to expand tissue for study device placement)
* Subject understands and signs the Informed Consent
* Subject agrees to return device to Mentor if device is explanted
* Subject agrees to comply with follow-up procedures, including returning for all follow-up visits
* Physician determines implant volume appropriate for the patient taking into account the subject's BMI and chest width

Exclusion Criteria:

* Subject is pregnant at time of enrollment
* Subject is a current smoker, or has smoked within 3 months prior to enrollment, or plans to resume smoking within 3 months post-enrollment
* Currently has uncontrolled diabetes (at time of screening or enrollment)
* Has nursed a child within 3 months of study enrollment
* Confirmed or suspected diagnosis of the following rheumatological autoimmune diseases or immune compromised status: SLE, Sjogren's syndrome, scleroderma, polymyositis, or any connective tissue disorder, rheumatoid arthritis, crystalline arthritis, infectious arthritis, spondyloarthropathies, any other inflammatory arthritis, fibromyalgia, or chronic fatigue syndrome
* Currently has a condition that could compromise or complicate wound healing. Note, obesity alone is not an exclusion. All surgical risk factors (obesity, diabetes, smoking history, and prior radiation) should be considered in totality for proper subject selection
* Infection or abscess anywhere in the body
* Demonstrates tissue characteristics that are clinically incompatible with successful use of a breast implant (e.g. inadequate tissue or compromised vascularity)
* Possesses any condition, or is under treatment for any condition which, in the opinion of the investigator and/or consulting physicians(s), may constitute an unwarranted surgical risk
* Anatomic or physiologic abnormality that could lead to significant postoperative adverse events
* Demonstrates characteristics that are unrealistic/unreasonable with the risks involved with the surgical procedure
* Untreated active, or inappropriately/inadequately treated breast malignancy, without surgical treatment
* Anticipated need for use of ADM/mesh at the time of implant or implant exchange
* Subject is HIV positive
* Works for Mentor or the study doctor or is directly related to anyone who works for Mentor or the study doctor
* Implanted metal or metal devices that make a MRI scan prohibitive, history of claustrophobia or other condition that would make a MRI scan prohibitive

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
10 Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Any Reoperation | 10 years
10 Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Baker III, IV Capsular Contracture | 10 year
10 Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Infection | 10 year
10 Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Explantation with or without replacement | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Mentor Worldwide, LLC
Locations (30):
- United States (30):
  - Plastic Surgery Associates of Montgomery, Montgomery, Alabama
  - Mosharrafa Plastic Surgery, Phoenix, Arizona
  - Mayo Clinic Arizona - Scottsdale/Phoenix (MCSB), Phoenix, Arizona
  - Andres Plastic Surgery, Scottsdale, Arizona
  - Adventist Health Bakersfield, Bakersfield, California
  - Susan E Downey MD, Inc, Burbank, California
  - Liu Plastic Surgery, Los Gatos, California
  - Stanford University School of Medicine, Stanford, California
  - Buckhead Plastic Surgery, P.C, Atlanta, Georgia
  - Georgia Institute of Plastic Surgery, Savannah, Georgia
  - The Centre, PC, Mishawaka, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - The University of Kansas, Kansas City, Kansas
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - The Mount Sinai Medical Center, New York, New York
  - Plastic Surgery Institute of Dayton, Centerville, Ohio
  - The Plastic Surgery Group, Cincinnati, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Plastic Surgery, Columbus, Ohio
  - Legacy Good Samaritan Medical Center, Portland, Oregon
  - Paul Glat, MD, PC, Bala-Cynwyd, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Center for Dermatology and Plastic Surgery at Springbrook, Alcoa, Tennessee
  - The Plastic Surgery Group PC, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Baylor Scott & White Health, Temple, Texas
  - UVA Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garvey PB, Larsen AN, Skoracki RJ, Djohan RS, Migliori MR, Tenenbaum MM, Friedman JD, Serletti JM, Rebecca AM, Kane WJ. Larger-volume Silicone Breast Implants Are Safe in Breast Reconstruction: the Athena Multicenter, Prospective Study of 400 Patients. Plast Reconstr Surg. 2026 Jan 22. doi: 10.1097/PRS.0000000000012840. Online ahead of print. PMID 41568948